CLINICAL TRIAL: NCT04682795
Title: A Prospective, Multi-center, Randomized, Open-label, Parallel Group Study to Evaluate Safety and Efficacy of Needle-free Injector Versus Insulin Pen in Patients With Type 2 Diabetes Mellitus
Brief Title: Comparison of Safety and Efficacy of Needle-Free Injector and Insulin Pen in Patients With T2DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-811
Record Dates: First submitted 2020-12-16; First posted 2020-12-24 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2020-12

CONDITIONS: T2DM (Type 2 Diabetes Mellitus); Needle-free Injector; Time in Range
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Needle-free injector group (Experimental): To evaluate the efficacy and safety of the needle-free injector in T2DM
  Interventions: Device: Needle-free injector
- Insulin pen group (Active Comparator): To evaluate the efficacy and safety of the insulin pen in T2DM
  Interventions: Device: Insulin pen

INTERVENTIONS:
Device: Needle-free injector — Using needle-free injector as insulin carrier to treat T2DM
  Arms: Needle-free injector group
Device: Insulin pen — Using insulin pen as insulin carrier to treat T2DM
  Arms: Insulin pen group

SUMMARY:
In this prospective, multi-center, randomized, open-label, parallel group trial, the safety and efficacy of needle-free injector will be compared with insulin pen after 2 weeks of treatment in patients with type 2 diabetes. This trial will enable assessment of the clinically relevant endpoint of a change in Time in Range (TIR), a newly recommended measurement of blood glucose fluctuations.

DETAILED DESCRIPTION:
The objective of the current study is to investigate the efficacy, safety and tolerability of needle-free injector compared to conventional insulin pen given for 2 weeks as the insulin carrier in patients with type 2 diabetes mellitus. The primary endpoint in this study is the change from baseline in TIR (after 2 weeks of treatment) in all patients with baseline and at least one post baseline measurement. Patients with type 2 diabetes who meet the entry criteria are planned for inclusion in this trial. Approximately 200 patients will be enrolled in the study. Patients who qualify will be randomized to needle-free injector group or conventional insulin pen group. Duration of treatment includes 1-week screening period, 2-week treatment observation period and 2-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 and ≤75 years with type 2 diabetes;
* HbA1c ≥ 7.5 to ≤11.0%;
* Receipt of premixed insulin and/or oral anti-diabetic agents ≥ 12 weeks before enrollment in the study, and insulin dose adjustments ≤ 10% within 4 weeks before enrollment (dose adjustment = (the maximum dose within a month - the minimum dose) / Final dose (dose of the day before the visit) × 100%);
* BMI ≤ 32kg / m2.

Exclusion Criteria:

* Patients with any of the following conditions will be excluded:
* Pregnant or lactating women
* Severe hypoglycemia within one month; diabetic ketoacidosis or hyperosmotic diabetic status within 6 months prior to informed consent
* Myocardial infarction, stroke or other severe cardiovascular events within 6 months prior to informed consent
* Current treatment with systemic steroids or immunosuppressive agents, or have immunologic deficiency disease at time of informed consent
* Severe mental instability, or alcohol abuse, or drug abuse
* Skin lesions at the insulin injection site
* Cancer within 5 years prior to informed consent
* Pancreatitis of severe infectious diseases within 1 months prior to informed consent
* Known hypersensitivity or allergy to the insulin
* Renal impairment (CKD-EPI eGFR<60ml/min)
* Impaired hepatic function, defined by serum levels of either ALT (SGPT), AST (SGOT), or alkaline phosphatase above 3 x upper limit of normal (ULN) as determined
* Participation in another trial within 2 months prior to informed consent
* Patients that investigators believe may fail to complete the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Time In Range | 2 weeks
  Time In Range (TIR, 3.9-10mmol/L)

SECONDARY OUTCOMES:
Time to occurrence of treat to target | 2 weeks
  Fasting glucose on treatment <7mmol/L and non-fasting glucose <10mmol/L, or TIR >70% (SMBG or FCGM)
Occurrence of a treat to target response and without any hypoglycemic episodes | 2 weeks
  Occurrence of a treat to target response and without any hypoglycemic episodes
EQ-5D Health Questionnaire | 2 weeks
  the EQ-5D descriptive system The change from baseline after 2 weeks of treatment
EQ-VAS Health Questionnaire | 2 weeks
  the EQ-VAS. The change from baseline after 2 weeks of treatment
Short Form 36 (SF-36) | 2 weeks
  The change from baseline after 2 weeks of treatment
Insulin dose | 2 weeks
  The change from baseline after 2 weeks of treatment

OTHER OUTCOMES:
Insulin treatment compliance | 2 weeks
  Recording whether the subjects obey the program to inject insulin at the specified time point in the 1st, 2nd, 3rd visit. Compliance will be calculated according to the formula: Compliance(%) = （Number of injections actually administered /Number of injections which should have been administered in the same period）*100%

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Changxing Campus, Changxing, Zhejiang
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang
  - 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Affiliated Hangzhou First People's Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The 2nd Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang
  - The First People's Hospital of Xiaoshan, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - Jinhua Municipal Central Hospital Medical Group, Jinhua, Zhejiang
  - Lanxi People's Hospital, Lanxi, Zhejiang
  - Lishui People's Hospital, Lishui, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - The Affiliated People's Hospital of Ningbo University, Ningbo, Zhejiang
  - Quzhou People's Hospital, Quzhou, Zhejiang
  - Shangyu People's Hospital of Shaoxing, Shaoxing, Zhejiang
  - The Affiliated Hospital of Shaoxing University, Shaoxing, Zhejiang
  - Taizhou Hospital, Taizhou, Zhejiang
  - Tongxiang First Hospital, Tongxiang, Zhejiang
  - The First People's Hospital of Wenling, Wenling, Zhejiang
  - Zhoushan Hospital, Zhoushan, Zhejiang

IPD SHARING:
Plan to Share IPD: No